CLINICAL TRIAL: NCT05963490
Title: A Prospective, Randomized, Controlled Phase II Trial of Regorafenib Alone or in Combination With Hypofractionated/Low-dose Radiotherapy Plus Toripalimab as Third-line Treatment in Patients With Metastatic Colorectal Cancer
Brief Title: Regorafenib Alone or in Combination With Hypofractionated/Low-dose Radiotherapy Plus Toripalimab for Metastatic Colorectal Cancer
Acronym: SLOT
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Zhen Zhang, Professor, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FDRT-2023-118-3237
Record Dates: First submitted 2023-07-19; First posted 2023-07-27 (Actual); Last update posted 2024-09-24 (Actual); Status verified 2024-09

CONDITIONS: Microsatellite Stable Metastatic Colorectal Cancer
MeSH Terms: interventions — regorafenib; toripalimab; Radiotherapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- monotherapy (Active Comparator): a total of 54 patients will receive regorafenib monotherapy.
  Interventions: Drug: Regorafenib
- combination therapies (Experimental): a total of 54 patients will first receive 1 cycle of regorafenib and toripalimab followed by hypofractionated/low-dose radiotherapy. Regorafenib and toripalimab will be continued after the completion of radiotherapy.
  Interventions: Drug: Toripalimab; Radiation: Radiotherapy; Drug: Regorafenib

INTERVENTIONS:
Drug: Regorafenib — Regorafenib 120 mg orally once daily on days 1-21 of each 28 days cycle.
  Other Names: Stivarga
  Arms: monotherapy
Drug: Toripalimab — 240 mg intravenously every 3 weeks
  Arms: combination therapies
Radiation: Radiotherapy — hypofractionated radiotherapy (5 fractions of 4-12Gy) and low-dose radiotherapy (5 fractions of 0.5-2Gy).
  Arms: combination therapies
Drug: Regorafenib — Regorafenib 80mg orally once daily on days 1-21 of each 28 days cycle.
  Arms: combination therapies

SUMMARY:
The study compares the efficacy and safety of regorafenib alone or in combination with hypofractionated radiotherapy and low-dose radiotherapy (LDRT) plus toripalimab in patients with microsatellite stable metastatic colorectal cancer (MSS mCRC). Patients are randomly assigned (1:1) into the control arm and the experimental arm. Control arm: a total of 54 patients will receive regorafenib monotherapy. Experimental arm: a total of 54 patients will first receive 1 cycle of regorafenib and toripalimab followed by hypofractionated/low-dose radiotherapy. Regorafenib and toripalimab will be continued after the completion of radiotherapy. The survival benefits, response rates, and adverse effects will be analyzed.

DETAILED DESCRIPTION:
Control arm: regorafenib 120 mg orally once daily on days 1-21 of each 28 days cycle.

Experimental arm: regorafenib is administered 80 mg once daily on days 1-21 of each 28 days cycle with intravenous toripalimab 240 mg every 3 weeks. Radiotherapy regimes include hypofractionated radiotherapy (5 fractions of 4-12Gy) and low-dose radiotherapy (5 fractions of 0.5-2Gy).

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years old
2. An Eastern Cooperative Oncology Group (ECOG) performance status ≤1
3. Life expectancy of at least 3 months
4. Histopathological confirmed MSS/pMMR adenocarcinoma of the colon or rectum
5. At least one evaluable metastatic lesion for radiotherapy according to RECIST 1.1
6. Progressed on or after the standard first-and second-line therapies or stopped standard therapy because of unacceptable toxic effects
7. Previous radiotherapy completed at least 4 weeks before randomization
8. Adequate bone-marrow, hepatic, and renal function: neutrophils ≥ 1.5 × 10^9/L, Hb ≥ 90 g/L, PLT ≥ 100 × 10^9/L, ALT/ AST≤2.5 ULN, Cr≤1 ULN
9. Sign the informed consent and have good compliance

Exclusion Criteria:

1. History of previous treatment with regorafenib and ICIs such as anti-PD-1 or anti-PD-L1 mAbs
2. Current severe cardiovascular diseases such as unstable angina, congestive heart failure, or serious cardiac arrhythmia requiring medication
3. Acute cardiac infarction or cerebral ischemic stroke occurred within 6 months before recruitment
4. Active autoimmune diseases and immunodeficiencies, known history of organ transplantation, or systematic use of immunosuppressive agents
5. Active Hepatitis B virus (HBV) or hepatitis C virus (HCV) infection: HBsAg positive or HBV DNA positive, anti-HCV antibody testing positive and confirmatory HCV RNA positive
6. Positive human immunodeficiency virus (HIV) infection, active syphilis infection, or active pulmonary tuberculosis infection
7. Severe infections requiring systemic antibiotics, antifungal or antiviral therapy
8. Uncontrollable pleural effusion, pericardial effusion, or ascites
9. Other malignancies within 5 years before recruitment, except for non-melanoma skin cancer, superficial bladder cancer, cervical carcinoma in situ, or breast cancer in situ that had been effectively treated.
10. Known history of severe neurological or mental illness such as schizophrenia, dementia, or epilepsy
11. Known history of allergy to any component involved in this study.
12. Pregnancy or breast-feeding women

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2023-04-25 (Actual); Primary Completion 2025-04-25 (Estimated); Study Completion 2026-04-25 (Estimated)

PRIMARY OUTCOMES:
OS | Up to 2 years
  Defined as the time from initiation of treatment to death from any cause.

SECONDARY OUTCOMES:
PFS | Up to 2 years
  Defined as the time from initiation of treatment to PD or death from any cause.
DCR | Up to 1 year
  The percentage of patients with disease control in all metastatic lesions. Disease control is defined as CR, PR, or stable disease (SD) per RECIST v1.1 and iRECIST after treatment.
ORR | Up to 1 year
  The percentage of patients with objective response in all metastatic lesions.
DoR | Up to 1 year
  Defined as the time between PR/CR and subsequent progression disease (PD) per RECIST v1.1 and iRECIST or death from any cause.
Adverse events | Up to 1 year
  The percentage of patients with treatment-related acute toxicities as assessed by NCI CTCAE v5.0, from treatment initiation until 90 days upon completion of immunotherapy.

CONTACTS AND LOCATIONS:
Overall Officials: Zhen Zhang, MD, PHD, Principal Investigator — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, China

REFERENCES:
- [Derived] Zhou S, Wang C, Shen L, Wang Y, Zhang H, Wu R, Wang Y, Chen Y, Xuan Y, Xia F, Zhang Z, Wan J. Regorafenib alone or in combination with high/low-dose radiotherapy plus toripalimab as third-line treatment in patients with metastatic colorectal cancer: protocol for a prospective, randomized, controlled phase II clinical trial (SLOT). Front Oncol. 2023 Oct 5;13:1274487. doi: 10.3389/fonc.2023.1274487. eCollection 2023. PMID 37869085